CLINICAL TRIAL: NCT06438965
Title: Multispectral Optoacoustic Imaging (MSOT) as Non-invasive Biomarker for Diagnosis and Monitoring of Neuromuscular Diseases (MSOT-NMD)
Brief Title: MSOT as Non-invasive Biomarker for Diagnosis and Monitoring of Neuromuscular Diseases
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Eastern Ontario (Other)
Responsible Party: Principal Investigator, Hanns Lochmuller, Professor of Neurology, Children's Hospital of Eastern Ontario
Other Study IDs: MSOT-01
Record Dates: First submitted 2024-05-10; First posted 2024-06-03 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Neuromuscular Diseases
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patient with neuromuscular disease: Muscle regions of the patients with neuromuscular diseases will be imaged using the MSOT device. Repeated measurements will be done after 6-12 months.
  Interventions: Device: Multispectral Optoacoustic Tomography (MSOT)

INTERVENTIONS:
Device: Multispectral Optoacoustic Tomography (MSOT) — MSOT scans will be obtained from two muscle region to measure hemo/myoglobin, collagen and lipid content/signal and oxygenation in patient with neuromuscular diseases.

SUMMARY:
The goal of this study is to learn if Multispectral Optoacoustic Tomographs (MSOT) works to diagnose and follow the course of neuromuscular diseases (NMDs) in children. MSOT scans will be obtained from muscle region to measure hemo/myoglobin, collagen and lipid content/signal and oxygenation in patients with neuromuscular diseases. No additional research activities -other than MSOT - will be done during this study. Existing clinical, laboratory and imaging data from standard-of-care procedures will be correlated with the MSOT data. The expected total duration of the study is approximately 36 months. Repeated measurements will be done to evaluate disease progression and the value of MSOT in NMD.

ELIGIBILITY:
Inclusion Criteria:

Patients with neuromuscular disease

* Children (from birth (infants that are born term) to 18 years of age) participants or consent through authorized guardian
* Confirmed or suspected diagnosis of a neuromuscular disease (through molecular genetics, biopsy, clinical examination)

Exclusion Criteria:

Participants:

* Diagnosis is not consistent with a confirmed or suspected neuromuscular disease
* Patients with active skin lesions (e.g. infections, trauma) or confirmed genetic disorders (e.g. epidermolysis bullosa) that predisposes to skin lesion
* Medically unstable patients
* Tattoo on skin overlying the area to be examined
* Missing consent form
* Exclusion due to safety concerns of the investigator (subject who has any condition, including any physical, psychological, or psychiatric condition, which in the opinion of the Investigator, would compromise the safety of the subject or the quality of the data and renders the subject an unsuitable candidate for the study)
* Medication leading to increased light sensitivity

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with various neuromuscular diseases who are seen at the Children's Hospital of Eastern Ontario will be offered to participate in the study as part of their diagnostic work-up and at regular intervals during their ongoing care.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2025-02-07 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Comparison of the quantitative proportion of collagen, lipid, and hemo/myoglobin signal | Every 6-12 month, assessed up to 36 months. Some people might be in the study for a very short time, some might be in it for 36 months depending on the time they join the study
  Comparison of the quantitative proportion of collagen, lipid, and hemo/myoglobin signal determined by MSOT in muscle tissue of patients with different neuromuscular diseases with their clinical data.

SECONDARY OUTCOMES:
Comparison of the quantitative amount of lipid and collagen signal | Every 6-12 month, assessed up to 36 months. Some people might be in the study for a very short time, some might be in it for 36 months depending on the time they join the study
  Comparison of the quantitative amount of lipid and collagen signal determined by MSOT in muscle tissue of children with different neuromuscular diseases.
Comparison of the quantitative proportion of oxygenated/deoxygenated hemo/myoglobin signal | Every 6-12 month, assessed up to 36 months. Some people might be in the study for a very short time, some might be in it for 36 months depending on the time they join the study
  Comparison of the quantitative proportion of oxygenated/deoxygenated hemo/myoglobin signal in muscle tissue of children with different neuromuscular diseases.
Comparison of the quantitative amount of oxygenated/deoxygenated hemo/myoglobin signal | Every 6-12 month, assessed up to 36 months. Some people might be in the study for a very short time, some might be in it for 36 months depending on the time they join the study
  Comparison of the quantitative amount of oxygenated/deoxygenated hemo/myoglobin signal determined by MSOT in muscle tissue of children with different neuromuscular diseases
Comparison of the MSOT-determined quantitative amount of hemo/myoglobin, lipid, and collagen signal at different positions /muscle groups intraindividually | Every 6-12 month, assessed up to 36 months. Some people might be in the study for a very short time, some might be in it for 36 months depending on the time they join the study
  Comparison of the MSOT-determined quantitative amount of hemo/myoglobin, lipid, and collagen signal at different positions /muscle groups intraindividually in children with different neuromuscular diseases, to identify disease specific distribution patterns
Comparison of the quantitative proportion of oxygenated/deoxygenated hemo/myoglobin, lipid, and collagen signal determined by MSOT at different positions /muscle groups intraindividually | Every 6-12 month, assessed up to 36 months. Some people might be in the study for a very short time, some might be in it for 36 months depending on the time they join the study
  Comparison of the quantitative proportion of oxygenated/deoxygenated hemo/myoglobin, lipid, and collagen signal determined by MSOT at different positions /muscle groups intraindividually in children with different neuromuscular diseases, to identify disease specific distribution patterns
Correlation of the collagen signal | Every 6-12 month, assessed up to 36 months. Some people might be in the study for a very short time, some might be in it for 36 months depending on the time they join the study
  Correlation of the collagen signal determined with MSOT with clinical assessments performed on a routine level during visits.
Correlation of the oxygenated/deoxygenated hemo/myoglobin signal determined with MSOT clinical assessments | Every 6-12 month, assessed up to 36 months. Some people might be in the study for a very short time, some might be in it for 36 months depending on the time they join the study
  Correlation of the oxygenated/deoxygenated hemo/myoglobin signal determined with MSOT clinical assessments performed on a routine level during visits.
Correlation of the collagen signal determined with MSOT with routine laboratory tests | Every 6-12 month, assessed up to 36 months. Some people might be in the study for a very short time, some might be in it for 36 months depending on the time they join the study
  Correlation of the collagen signal determined with MSOT with routine laboratory tests such as blood creatine kinase (CK) levels, transaminases.
Correlation of the oxygenated/deoxygenated hemo/myoglobin signal determined by MSOT with routine laboratory tests | Every 6-12 month, assessed up to 36 months. Some people might be in the study for a very short time, some might be in it for 36 months depending on the time they join the study
  Correlation of the oxygenated/deoxygenated hemo/myoglobin signal determined by MSOT with routine laboratory tests such as blood CK levels, transaminases.
Correlation of the collagen signal determined with MSOT with patient reported outcome measures. | Every 6-12 month, assessed up to 36 months. Some people might be in the study for a very short time, some might be in it for 36 months depending on the time they join the study
  Correlation of the collagen signal determined with MSOT with patient reported outcome measures.
Correlation of the oxygenated/deoxygenated hemo/myoglobin signal determined by MSOT with patient reported outcome measures. | Every 6-12 month, assessed up to 36 months. Some people might be in the study for a very short time, some might be in it for 36 months depending on the time they join the study
  Correlation of the oxygenated/deoxygenated hemo/myoglobin signal determined by MSOT with patient reported outcome measures.
Correlation of the collagen signal determined with MSOT with the current treatment regimen | Every 6-12 month, assessed up to 36 months. Some people might be in the study for a very short time, some might be in it for 36 months depending on the time they join the study
  Correlation of the collagen signal determined with MSOT with the current treatment regimen in patients with NMD.
Correlation of the oxygenated/deoxygenated hemo/myoglobin signal determined by MSOT with the current treatment regimen | Every 6-12 month, assessed up to 36 months. Some people might be in the study for a very short time, some might be in it for 36 months depending on the time they join the study
  Correlation of the oxygenated/deoxygenated hemo/myoglobin signal determined by MSOT with the current treatment regimen in patients with NMD.

CONTACTS AND LOCATIONS:
Locations (1):
- CHEO, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No